CLINICAL TRIAL: NCT00677300
Title: Evaluation of Safety and Efficacy of Raltegravir/Darunavir Combination in Antiretroviral-Naive Patients
Brief Title: Raltegravir And Darunavir Antiretroviral in Antiretroviral Naive Patients
Acronym: RADAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dallas VA Medical Center (U.S. Federal Agency)
Collaborators: Merck Sharp & Dohme LLC (Industry); Tibotec Pharmaceutical Limited (Industry)
Responsible Party: Principal Investigator, Roger Bedimo, M.D., ID Section Chief, Dallas VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Merck 072-00
Record Dates: First submitted 2008-05-08; First posted 2008-05-14 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: HIV Infections
Keywords: HIV; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium; Darunavir; Ritonavir; Tenofovir; Emtricitabine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Will receive Raltegravir (400mg twice daily) + Ritonavir-boosted (100mg once daily) Darunavir (800mg once daily)
  Interventions: Drug: Raltegravir; Drug: Darunavir; Drug: Ritonavir
- Group B (Active Comparator): Will receive Tenofovir (300mg once daily) + Emtricitabine (200mg once daily) + Ritonavir-boosted (100mg once daily) Darunavir (800mg once daily)
  Interventions: Drug: Darunavir; Drug: Ritonavir; Drug: Tenofovir/Emtricitabine

INTERVENTIONS:
Drug: Raltegravir — 400mg P.O. (orally) twice daily for 48 weeks
  Other Names: Isentris
  Arms: Group A
Drug: Darunavir — 800 mg P.O. (orally) once daily
  Other Names: Prezista
Drug: Ritonavir — 100mg once daily
  Other Names: Norvir
Drug: Tenofovir/Emtricitabine — 300 mg/200 mg P.O. (orally) once daily
  Other Names: Truvada
  Arms: Group B

SUMMARY:
The purpose of this study is to determine whether a combination of raltegravir and darunavir is as effective as standard regimens in the treatment of HIV-infected patients who have not previously used antiretroviral drug (treatment naive)

DETAILED DESCRIPTION:
STUDY RATIONALE:

The current guidelines for HIV treatment in antiretroviral naive patients recommend the use of two drugs in the nucleoside reverse transcriptase inhibitor (NRTI) class in addition to one drug in the protease inhibitor (PI) or in the non-nucleoside reverse transcriptase inhibitor (NNRTI) class.

NRTI use is associated with significant toxicity, including mitochondrial dysfunction (mostly attributed to thymidine-analogue NRTIs): lipoatrophy, peripheral neuropathy, pancreatitis, lactic acidosis. There's also a significant risk of hypersensitivity reaction from Abacavir, and caution is needed when using Tenofovir in patients with renal failure.

Finding effective NRTI-free regimens would have a number of potential benefits including: 1) a significant expansion of therapeutic options; despite the growing number of antiretrovirals, treatment options might still be significantly limited in a patient with a number of baseline NRTI mutations or poor NRTI tolerance; 2) potential avoidance of toxicities.

Raltegravir is a leading candidate in a new class of antiretroviral medications called integrase inhibitors. It is currently approved for use in antiretroviral treatment experienced patients, but has been shown to have excellent virologic efficacy in naïve as well as heavily treatment experienced patients. It also has been shown to have unusually rapid virologic response. This profile might be excellent in delaying emergence of viral resistance in naïve patients.

Three phase III trials of Raltegravir in treatment experienced patients have been conducted (BENCHMRK trials). In both of these studies, more than 75 percent of patients receiving Raltegravir plus optimized background therapy (OBT) achieved viral load (HIV RNA) reductions to less than 400 copies/mL compared to more than 40 percent of patients receiving placebo plus OBT. Both studies also showed that Raltegravir plus OBT was generally well tolerated.

Darunavir is currently approved for use in HAART-experienced patients at the dose of 600 mg bid with ritonavir boosting. In subgroup analysis of the BENCHMRK trials, use of Raltegravir and Darunavir was associated with 90% virologic responses (HIV RNA < 400 copies/mL) at 24 weeks in treatment experienced subjects. Also, the recently presented ARTEMIS study found once-daily Darunavir to be non-inferior to either once- or twice-daily lopinavir/ritonavir in antiretroviral naïve patients. After 48 weeks a time-to-loss-of-virologic response analysis determined that 84% assigned to darunavir and 78% assigned to lopinavir had a viral load below 50 copies. In subgroup analysis, DRV/r QD was superior to LPV/r (overall) in patients with baseline viral load ≥100,000 copies/mL Furthermore, the DRV/r QD group experienced a lower incidence of lipid abnormalities than the lopinavir/ritonavir group.

HYPOTHESES

We hypothesize that the virologic efficacy (time to loss of virologic response) at 48 weeks will be at least as high following a regimen of Raltegravir + boosted Darunavir as with a regimen of Tenofovir + Emtricitabine + boosted Darunavir.

We further hypothesize that a regimen of Raltegravir + boosted Darunavir will not result in higher rates of adverse events at 48 weeks than a regimen of Tenofovir + Emtricitabine + boosted Darunavir.

STUDY DESIGN AND DURATION

This is a randomized, active Control, safety/efficacy study. All eligible patients (antiretroviral naïve,) will be randomized (1:1) into two treatment groups:

1. Group A: will receive Raltegravir + Ritonavir-boosted Darunavir
2. Group B: will receive Tenofovir + Emtricitabine + Ritonavir-boosted Darunavir

ELIGIBILITY:
Inclusion Criteria

* The patient has documented HIV-1 infection.
* The patient is at least 18 years of age.
* Antiretroviral naive, defined as 7 days or less of ARV treatment at any time prior to study entry. HIV viral load greater than 5,000 copies/ml within 90 days of study entry
* Willing to use acceptable forms of contraception
* Parent or guardian willing to provide informed consent, if applicable
* Hepatitis B surface antigen (HBsAg) negative at study entry

Exclusion Criteria

* Patient is current participant in a Raltegravir trial or in trials involving any of the other study medications (Darunavir, Tenofovir or Emtricitabine).
* Immunomodulators (e.g., interleukins, interferons, cyclosporine), HIV vaccine, systemic cytotoxic chemotherapy, or investigational therapy within 30 days prior to study entry. Individuals receiving either stable physiologic glucocorticoid doses, corticosteroids for acute therapy for pneumocystis pneumonia, or a short course (2 weeks or less) of pharmacologic glucocorticoid therapy will not be excluded.
* Known allergy/sensitivity to study drugs or their formulations
* Patient has a condition (including but not limited to active alcohol or drug use) that, in the opinion of the investigator, may interfere with patient adherence or safety
* Patient with acute hepatitis due to any cause or clinically significant chronic liver disease including but not limited to cirrhosis, ascites, encephalopathy, hypoalbuminemia, prolonged PT/PTT and/or esophageal varices.
* Patient has severe renal insufficiency defined as a calculated creatinine clearance at time of screening <30 mL/min, base on Cockcroft/Gault equation which is as follows (and 0.85 X this value for females):
* CrCl (mL/min) = [(140-Age) x Weight (in Kg)]/72 x Serum Creatinine (mg/mL)
* Serious illness requiring systemic treatment or hospitalization. Patients who have completed therapy or are clinically stable on therapy for at least 7 days prior to study entry are not excluded.
* Known clinically relevant cardiac conduction system disease
* Patient requires or is anticipated to require any of the prohibited medications noted in the protocol
* Current imprisonment or involuntary incarceration for psychiatric or physical (e.g., infectious disease) illness
* Pregnancy and Breastfeeding. Women who become pregnant during the study will be required to permanently discontinue their study regimens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2009-01; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Time from randomization to virologic failure (HIV viral load of 1,000 copies/ml or greater at or after Week 16 and before Week 24, or two consecutive HIV viral load of 50 copies/ml or greater at or after Week 24) | Week 24

SECONDARY OUTCOMES:
Median change in CD4 count from baseline | 48 Weeks
Percentage of patients with treatment-emergent fasting hypertriglyceridemia (TG >400) or hypercholesterolemia (TC >240) | 48 weeks
Median change in limb fat from baseline, by DEXA scan | 48 weeks
Changes from baseline in insulin resistance measured by homeostasis model assessment (HOMA-IR) | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roger Bedimo, M.D., Principal Investigator — Dallas VA Medical Center
Locations (2):
- United States (2):
  - Dallas VA Medical Center, Dallas, Texas
  - Parkland Health & Hospital System, Dallas, Texas

REFERENCES:
- [Derived] Bedimo RJ, Drechsler H, Jain M, Cutrell J, Zhang S, Li X, Farukhi I, Castanon R, Tebas P, Maalouf NM. The RADAR study: week 48 safety and efficacy of RAltegravir combined with boosted DARunavir compared to tenofovir/emtricitabine combined with boosted darunavir in antiretroviral-naive patients. Impact on bone health. PLoS One. 2014 Aug 29;9(8):e106221. doi: 10.1371/journal.pone.0106221. eCollection 2014. PMID 25170938